CLINICAL TRIAL: NCT07136792
Title: Efficacy and Safety of Pegmolesatide in Dialysis Chronic Kidney Disease (CKD) Patients With Anemia Treated With Hypoxia-inducible Factor Prolyl Hydroxylase Inhibitor (HIF-PHI): a Multi-center, Prospective, Open-label, Randomized Parallel Controlled Trial
Brief Title: A Study of Pegmolesatide of in Dialysis Chronic Kidney Disease (CKD) Patients With Anemia Treated With Hypoxia-inducible Factor Prolyl Hydroxylase Inhibitor (HIF-PHI)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Guangdong Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, XueQing Yu, professor, Guangdong Provincial People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KY2025-667-03
Record Dates: First submitted 2025-07-31; First posted 2025-08-22 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Renal Anemia of Chronic Kidney Disease
Keywords: Renal Anemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Arm A1: Pegmolesatide 2mg SC (Experimental): All patients in low-dose Roxadustat cohort randomised into this group will receive pegmolesatide 2mg subcutaneously once every 4 weeks.
  Interventions: Drug: Pegmolesatide 2mg SC
- Arm A2: Pegmolesatide 4mg SC (Experimental): All patients in low-dose Roxadustat cohort randomised into this group will receive pegmolesatide 4mg subcutaneously once every 4 weeks.
  Interventions: Drug: Pegmolesatide 4mg SC
- Arm B1: Pegmolesatide 4mg SC (Experimental): All patients in high-dose Roxadustat cohort randomised into this group will receive pegmolesatide 4mg subcutaneously once every 4 weeks.
  Interventions: Drug: Pegmolesatide 4mg SC
- Arm B2: Pegmolesatide 6mg SC (Experimental): All patients in high-dose Roxadustat cohort randomised into this group will receive pegmolesatide 6mg subcutaneously once every 4 weeks.
  Interventions: Drug: Pegmolesatide 6mg SC

INTERVENTIONS:
Drug: Pegmolesatide 2mg SC — All patients will receive pegmolesatide 2mg subcutaneously once every 4 weeks.
  Arms: Arm A1: Pegmolesatide 2mg SC
Drug: Pegmolesatide 4mg SC — All patients will receive pegmolesatide 4mg subcutaneously once every 4 weeks.
  Arms: Arm A2: Pegmolesatide 4mg SC
Drug: Pegmolesatide 4mg SC — All patients will receive pegmolesatide 4mg subcutaneously once every 4 weeks.
  Arms: Arm B1: Pegmolesatide 4mg SC
Drug: Pegmolesatide 6mg SC — All patients will receive pegmolesatide 6mg subcutaneously once every 4 weeks.
  Arms: Arm B2: Pegmolesatide 6mg SC

SUMMARY:
For patients with renal anemia treated with hypoxia-inducible factor prolyl hydroxylase inhibitor (HIF-PHI), there is a clinical need of switching to long-acting and safe medications.

Pegmolesatide, a polyethylene glycol (PEG)-conjugated erythropoiesis-stimulating peptide, is a long-acting erythropoiesis-stimulating agent (ESA) with sustained activity. It was approved for marketing by the National Medical Products Administration (NMPA) in June 2023. Phase III clinical trials have demonstrated its efficacy and safety in dialysis patients with renal anemia who were previously treated with recombinant human erythropoietin (rHuEPO). However, there are currently no data regarding the efficacy and safety of switching from HIF-PHIs to pegmolesatide, and there is a lack of standard for the dose conversion.

This study is a multi-center, prospective, open-label, randomized parallel-controlled clinical trial, planning to enroll 96 patients.

All enrolled patients will receive 12 weeks of treatment and be followed up for 16 weeks.

DETAILED DESCRIPTION:
For patients with renal anemia treated with HIF-PHIs, there is a clinical need of switching to long-acting and safe medications.

Pegmolesatide, a polyethylene glycol (PEG)-conjugated erythropoiesis-stimulating peptide, is a long-acting erythropoiesis-stimulating agent (ESA) with sustained activity. It was approved for marketing by the National Medical Products Administration (NMPA) in June 2023. Phase III clinical trials have demonstrated its efficacy and safety in dialysis patients with renal anemia who were previously treated with recombinant human erythropoietin (rHuEPO). However, there are currently no data regarding the efficacy and safety of switching from HIF-PHIs to pegmolesatide, and there is a lack of standard for the dose conversion.

This study is a multi-center, prospective, open-label, randomized parallel-controlled clinical trial, planning to enroll 96 patients.

Based on the weekly dose of Roxadustat before randomization, patients are divided into two cohorts: the low-dose Roxadustat cohort (weekly dose ≤210 mg) and the high-dose Roxadustat cohort (weekly dose >210 mg and ≤360 mg), with 48 patients in each cohort. Each cohort is stratified by hemoglobin (HB) level, with a 1:1 ratio for HB <10.0 g/dl and HB ≥10.0 g/dl, meaning that there are 24 patients in both cohorts.

Within each cohort, patients are randomly assigned to 2 groups at a 1:1 ratio based on the initial treatment dose of pegmolesatide. Specifically, the patients in low-dose Roxadustat cohort are randomized into the Pegmolesatide initial dose 2 mg group or 4 mg group; the patients in high-dose Roxadustat cohort are randomized into the Pegmolesatide initial dose 4 mg group or 6 mg group, with 24 patients in each group entering the trial period. Pegmolesatide is administered subcutaneously once every 4 weeks, and the dosage is adjusted according to the drug's instructions for use. All enrolled patients will receive 12 weeks of treatment and be followed up for 16 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18-75 years, regardless of gender;
2. Body weight ≥ 45 kg, and body mass index (BMI) ≥ 18.5 kg/m²;
3. Diagnosis of chronic renal failure, and having undergone a stable regimen of peritoneal dialysis or hemodialysis for at least 12 weeks prior to enrollment (with stable hemofiltration at a frequency of every 2 or 4 weeks if applicable). Stable dialysis frequency and no plans to change the dialysis modality during the trial;
4. An up to standard dialysis adequacy testing result before randomization: spKt/V ≥ 1.2 for hemodialysis, Kt/V ≥ 1.7 for peritoneal dialysis;
5. Roxadustat dose ≤ 360 mg/week within 4 weeks before randomization, with stable dose; [Stable dose is defined as: (the maximum weekly dose within 4 weeks before randomization - the average weekly dose within 4 weeks before randomization) ÷ the maximum weekly dose within 4 weeks before randomization ≤ 30%];
6. Two pre-dialysis HB test values within 4 weeks before randomization of 8.0 - 12.0 g/dl, with an absolute difference between the two Hb values ≤ 1.3 g/dl, and an interval of ≥ 7 days between the two HB tests;
7. Serum ferritin level ≥ 100 μg/L and transferrin saturation (TAST) ≥ 20% at the time of testing before randomization, serum folate ≥ the lower limit of normal, and vitamin B12 ≥ the lower limit of normal;
8. Understanding of the study procedures and voluntary signing of the written informed consent form.

Exclusion Criteria:

1. Known autoimmune diseases, hematologic disorders (including congenital and acquired conditions such as thalassemia, Fanconi anemia, pure red cell aplasia, myelodysplastic syndrome, hemolytic anemia, and coagulation disorders), or other causes of anemia apart from CKD (such as gastrointestinal bleeding or hookworm disease).
2. Confirmed diagnosis of acquired immunodeficiency syndrome (AIDS), syphilis, or tuberculosis and currently undergoing treatment.
3. Known allergy to iron agents or polyethylene glycol molecules.
4. Treatment history with ESAs in combination with HIF-PHIs drugs within 8 weeks prior to randomization.
5. Underwent red blood cell or whole blood transfusion within 12 weeks prior to randomization.
6. Poorly controlled blood pressure (uncontrolled hypertension is defined as: during the screening period, systolic blood pressure > 180 mmHg or diastolic blood pressure > 110 mmHg in two or more blood pressure measurements, or although the blood pressure values are below the aforementioned criteria, the investigator deems it necessary to adjust antihypertensive medications).
7. Active hepatitis or any of the following abnormal test results during the screening period (ALT ≥ 2 times the upper limit of normal, AST ≥ 2 times the upper limit of normal, DBIL ≥ 2 times the upper limit of normal, serum albumin < 2.5 g/dl).
8. Participants judged by the investigator to have uncontrolled or symptomatic secondary hyperparathyroidism, or those with blood iPTH > 800 pg/mL during the screening period.
9. C-reactive protein ≥ 30 mg/L during the screening period.
10. Cardiac function assessed as NYHA Class III or IV during the screening period.
11. Pregnant or breastfeeding women, or those planning to become pregnant during the study period.
12. Participants who plan to undergo kidney transplantation during the trial period or have already been kidney donors, or those who plan to undergo elective surgery during the trial period.
13. Participants deemed by the investigator to have any other factors that make them unsuitable for participation in this trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2025-09-08 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Change of mean HB level | from baseline to 12 weeks and 16 weeks
  Change of mean HB level from baseline to 12 weeks and 16 weeks

SECONDARY OUTCOMES:
Change of mean HB level | from baseline to 12 weeks and 16 weeks
  Change in mean HB levels from baseline to 12 weeks and 16 weeks, stratified by different baseline HB levels
Changes in red blood cell count | from baseline to 4 weeks, 8 weeks, 12 weeks, 16 weeks
  Changes in red blood cell count from baseline to each follow-up
Median time to the first HB value reaching 10.0-12.0 g/dl | From baseline to 4 weeks, 8 weeks,12 weeks and 16 weeks
  Median time to the first HB value reaching 10.0-12.0 g/dl
Proportion of patients with HB 10.0-12.0 g/dl | from baseline to 4 weeks, 8 weeks,12 weeks and 16 weeks
  Proportion of patients with HB 10.0-12.0 g/dl at each follow-up
Proportion of patients with HB 11.0-13.0 g/dl | from baseline to 4 weeks, 8 weeks, 12 weeks and 16 weeks
  Proportion of patients with HB11.0-13.0 g/dl at each follow-up
Average drug dose at each follow-up | From baseline to 4 weeks, 8 weeks,12 weeks and 16 weeks
Adverse Events | From the start of study drug to 30 days after the last dose of study drug
  Safety of therapy by Investigator.

OTHER OUTCOMES:
The Maximum Plasma Concentration | from the start of study drug to to 48 hours, 72 hours and 96 hours
  The Maximum Plasma Concentration of Pegmolesatide

CONTACTS AND LOCATIONS:
Overall Officials: Xueqing Yu, Study Chair — Guangdong Provincial People's Hospital; Zhiming Ye, Study Director — Guangdong Provincial People's Hospital
Locations (24):
- China (24):
  - Beijing Hospital, Beijing, Beijing Municipality
  - Longyan First Hospital, Longyan, Fujian
  - Zhangzhou Municipal Hospital of Fujian Province, Zhangzhou, Fujian
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - Meizhou People's Hospital, Meizhou, Guangdong
  - The First Affiliated Hospital of Shantou University Medical College, Shantou, Guangdong
  - Yuebei People's Hospital, Shaoguan, Guangdong
  - Zhongshan Hospital of Traditional Chinese Medicine, Zhongshan, Guangdong
  - Affiliated Hospital of Zunyi Medical University, Zunyi, Guizhou
  - Jingmen Central Hospital, Jingmen, Hubei
  - CNPG Dongfeng General Hospital, Shiyan, Hubei
  - Tongji Hospital Affiliated to Tongji Medical College of Huazhong University of Science and Technology, Wuhan, Hubei
  - Wuhan Fourth Hospital, Wuhan, Hubei
  - Changsha Central Hospital, Changsha, Hunan
  - Nantong First People's Hospital, Nantong, Jiangsu
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - The First Affiliated Hospital of Baotou Medical College, Baotou, Neimenggu
  - The First Affiliated Hospital of Shandong First Medical University, Jinan, Shandong
  - Yibin First People's Hospital, Yibin, Sichuan
  - Tianjin First Center Hospital, Tianjin, Tianjin Municipality
  - Hangzhou Xiaoshan First People's Hospital, Hangzhou, Zhejiang
  - The Affiliated People's Hospital of Ningbo University, Ningbo, Zhejiang
  - Rui'an People's Hospital, Wenzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No